CLINICAL TRIAL: NCT03338868
Title: Comparison of Serum Concentrations, Physical and Psychological Well-being in Patients Having Chronic Musculoskeletal Pain With and Without Metabolic Syndrome
Brief Title: Serum Concentrations, Physical and Psychological Well-being in Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, PT, PhD, Ataturk Training and Research Hospital
Other Study IDs: 2015-13/32
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Metabolic Syndrome
Keywords: physical activity; pain; uric acid
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Pain | interventions — Body Composition; Quality of Life; Mental Health; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MetS: To be a volunteer patient with a chronic non-specific musculoskeletal pain disorder, including knee osteoarthritis, rotator cuff tear, adhesive capsulitis, and non-specific low back, back or neck pain for more than 6 months.
  Interventions: Other: Body composition; Other: Physical activity level; Other: Musculoskeletal pain intensity; Other: Quality of life; Other: Psychological Well-Being; Diagnostic Test: Blood tests
- Patients without MetS: To be a volunteer patient with a chronic non-specific musculoskeletal pain disorder, including knee osteoarthritis, rotator cuff tear, adhesive capsulitis, and non-specific low back, back or neck pain for more than 6 months.
  Interventions: Other: Body composition; Other: Physical activity level; Other: Musculoskeletal pain intensity; Other: Quality of life; Other: Psychological Well-Being; Diagnostic Test: Blood tests

INTERVENTIONS:
Other: Body composition — evaluated by Bodystat®1500 Bio-impedance Analyzer
Other: Physical activity level — assessed by the International Physical Activity Questionnaire-7
Other: Musculoskeletal pain intensity — evaluated with Visual Analog Scale
Other: Quality of life — assessed by the Nottingham Health Profile
Other: Psychological Well-Being — assessed by the Hospital Anxiety and Depression Scale
Diagnostic Test: Blood tests — Blood tests included serum glucose, triglyceride, high-density lipoprotein cholesterol (HDL-C), and uric acid levels. Blood samples were collected from the patients after one night of fasting.

SUMMARY:
The purpose of this study was to investigate the serum concentrations, physical and psychological well-being characteristics in patients having chronic musculoskeletal pain with metabolic syndrome, and to compare patients without metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a combination of metabolic risk factors such as impaired glucose level, dyslipidemia, hypertension, and central obesity. MetS has become a large public health issue with common interrelation to different accompanying disorders. Moreover, the link between MetS and musculoskeletal disorders has previously been demonstrated.

Presence and prevalence of MetS in patients having musculoskeletal pain seems common and interrelated.However, to our knowledge, manifestations with clinical symptoms of MetS, some inflammatory markers via serum concentrations and physical and psychological health profiles of patients with seeking treatment from outpatient physical therapy for musculoskeletal pain conditions have not been researched up to now.

ELIGIBILITY:
Inclusion Criteria:

To be a volunteer patient with a chronic non-specific musculoskeletal pain disorder, including knee osteoarthritis, rotator cuff tear, adhesive capsulitis, and non-specific low back, back or neck pain for more than 6 months.

Exclusion Criteria:

the presence of severe physical disability, psychiatric disorder, malignant tumors, pregnancy, chronic alcohol consumption, gout, heart failure, liver and renal dysfunction.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having chronic musculoskeletal pain with and without metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood tests | 2 years
  for uric acid levels.

SECONDARY OUTCOMES:
Body composition | 2 years
  evaluated by Bodystat®1500 Bio-impedance Analyzer
Physical activity level | 2 years
  assessed by the International Physical Activity Questionnaire-7. The intensity of self-reported physical activity, lasting at ten minutes per bout, was used to assess metabolic equivalent (MET). The MET is defined as the ratio of a working metabolic rate to a standard resting metabolic rate.MET-minutes/week was computed by multiplying the MET score of an activity (3.3 for walking, 4.0 for moderate-intensity, and 8.0 for vigorous-intensity) by the minutes and days performed. The summation of walking, moderate, and vigorous METs-minutes/week enabled the computation of the total physical activity performed by an individual.
The musculoskeletal pain intensity | 2 years
  evaluated with 0 to 10 cm Visual Analog Scale. "0" indicated "no pain" and the "10" indicated "the worst imaginable pain".
Quality of life | 2 years
  evaluated with the Nottingham Health Profile (NHP). It contains 38 items divided into 6 dimensions: NHP-energy, NHP-pain, NHP-emotional reactions, NHP sleep, NHP-social isolation, and NHP-physical mobility. All the parameters are summed as NHP-total. The respondent answers "yes" if the statement adequately reflected the current status or feeling, or "no" otherwise. Dimension scores ranged from 0 (no problems) to 100 (maximum problems).
Psychological Well-Being (Anxiety and Deppression condition) | 2 years
  evaluated with the Hospital Anxiety and Depression Scale (HADS). Each question was scored on a 4-point Likert scale, ranging from 0 to 3, where a higher score represented more severe anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Assist prof, Study Director — Ankara Yildirim Beyazit University Ataturk Training and Research Hospital
Locations (1):
- Ataturk Training and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Afzal N, Mahmud TE, Jahan SS, Kundi S. Uric acid profile in patients with chronic nonspecific musculoskeletal pain. J Ayub Med Coll Abbottabad. 2003 Oct-Dec;15(4):5-9. PMID 15067822
- [Result] Fu YQ, Yang H, Zheng JS, Zeng XY, Zeng W, Fan ZF, Chen M, Wang L, Li D. Positive association between metabolic syndrome and serum uric acid in Wuhan. Asia Pac J Clin Nutr. 2017 Mar;26(2):343-350. doi: 10.6133/apjcn.012016.06. PMID 28244715
- [Result] Chu AH, Moy FM. Association between physical activity and metabolic syndrome among Malay adults in a developing country, Malaysia. J Sci Med Sport. 2014 Mar;17(2):195-200. doi: 10.1016/j.jsams.2013.04.003. Epub 2013 May 9. PMID 23665093
- [Result] Saboya PP, Bodanese LC, Zimmermann PR, Gustavo AD, Assumpcao CM, Londero F. Metabolic syndrome and quality of life: a systematic review. Rev Lat Am Enfermagem. 2016 Nov 28;24:e2848. doi: 10.1590/1518-8345.1573.2848. PMID 27901223
- [Result] Takeuchi T, Nakao M, Nomura K, Inoue M, Tsurugano S, Shinozaki Y, Yano E. Association of the metabolic syndrome with depression and anxiety in Japanese men: a 1-year cohort study. Diabetes Metab Res Rev. 2009 Nov;25(8):762-7. doi: 10.1002/dmrr.1041. PMID 19839027